CLINICAL TRIAL: NCT05833464
Title: Cost-effectiveness Pharmacoeconomic Study of a Standardized Multidisciplinary Weight Loss Method (PronoKal® Method) to Improve the Health Condition of Obese Patients With Associated Comorbidities
Brief Title: Cost-effectiveness Study of a Multidisciplinary Weight Loss Method to Improve the Health Condition of Obese Patients
Acronym: PRONOCOST
Status: Withdrawn | Type: Observational
Why Stopped: The study was not started and no patients were recruited because the weight loss program was no longer prescribed in Argentina (the country where the study was to be carried out).
Sponsor: Protein Supplies SL (Other)
Responsible Party: Sponsor
Other Study IDs: PRO-COST-2016-02
Record Dates: First submitted 2018-05-08; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Obese
Keywords: comorbidities; PronoKal® Method; Cost-Benefit Analysis; loss weight; obesity
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational, multicenter study based on a registry of patients with obesity and associated comorbidities undergoing a standardized multidisciplinary weight loss method with a 2-year follow-up.

DETAILED DESCRIPTION:
The investigators will include obese patients with BMI higher than 30 kg / m2 and one or more comorbidities associated with obesity who are following a standardized multidisciplinary weight-loss program (PronoKal® Method), which consists of a very-low-calorie diet, into which natural foods are gradually reintroduced, accompanied by physical exercise and emotional support.

The aim of this study is to assess the cost-effectiveness to improve the health condition of obese patients with comorbidities and thereby reduce healthcare expenditure (pharmacological treatment, incidence of complications, use of health resources) and work absenteeism.

Patients will be monitored for 2 years. The registry of patient data for this study will be made by the doctor and dietitians / nutritionists who will regularly see the patient in the face-to-face visits at the Pronokal center.

The study will begin with the baseline visit (day 0) in which the inclusion and exclusion criteria will be confirmed, the signing of informed consent will be obtained and the multidisciplinary treatment will be prescribed, followed by 6 control visits: 2 visits during the ketogenic stage (1-month after the start and at the end of ketosis), 2 visits during the physiological adaptation phase (at 4 or 5 months and at the end of stage 2) and 2 follow-up visits during the maintenance up to the 2-year completion.

Likewise, dietitians/nutritionists, according to the methodology of the program, will carry out a face-to-face follow-up of the patient, which will be fortnightly during the ketogenic diet, monthly during the physiological adaptation of stage 2 and quarterly or semi-annual during the maintenance stage.

The information about the endpoints will be collected:

* Costs of weight loss treatment: products and dietary supplements + number of control visits + number of laboratory tests performed
* Healthcare expenditure: pharmacological treatment of associated comorbidities, incidence of complications (visits to his/her primary care physician, a specialist or emergency department for acute complications, treatment of acute complications, number of hospital admission days, antibiotic treatment), consumption of health resources (visits to the general practitioner, visits to specialists, laboratory tests)
* Work absenteeism: number of work leave days + hours of work absenteeism due to health problems or medical visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes 18 years of age or older
* Patients with overweight or obesity (BMI> 30 kg/m2) with at least one or more of the following comorbidities associated with obesity (type 2 diabetes mellitus, arterial hypertension, dyslipidemia, hyperuricemia) those who are under pharmacological treatment with two or more drugs (oral antidiabetic and/or lipid-lowering agents and/or antihypertensive and/or hypouricemic agents)
* Patients who agree to attend the follow-up visits at the Pronokal centre, in Buenos Aires.
* Patients who agree to participate and provide a signed informed consent

Exclusion Criteria:

* Patients who do not sign the informed consent
* Pregnant or breastfeeding patients.
* Patients with severe eating disorders, alcoholism, or substance abuse.
* Patients with severe psychological disorders (e.g., schizophrenia, bipolar disorder).
* Patients with liver failure.
* Patients with kidney failure.
* Patients with type 1 DM or insulin-dependent, or currently under insulin treatment, or candidates for insulin treatment in a short period of time.
* Patients with obesity caused by other endocrine diseases (except type 2 DM).
* Patients with blood disorders.
* Patients with cancer.
* Patients with cardiovascular or cerebrovascular disease (heart rhythm disorders, recent infarction [<6m], unstable angina, decompensated heart failure, recent stroke [<6m]).
* Patients with renal lithiasis.
* Patients with cholelithiasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients, with obesity-associated comorbidities, treated with the standardized multidisciplinary weight loss method (PronoKal® Method).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Healthcare expenditure for one year | 1 year
  Sum of the following costs: pharmacological treatment of associated comorbidities + visits to primary care physician + visits to specialist + visits to emergency department for acute complications +treatment for acute complications +number of hospital admission days + antibiotic treatment +laboratory tests, for one year (from baseline to 1 year)

SECONDARY OUTCOMES:
Healthcare expenditure the second year | 2 years
  Sum of the following costs: pharmacological treatment of associated comorbidities + visits to primary care physician + visits to specialist + visits to emergency department for acute complications +treatment for acute complications +number of hospital admission days + antibiotic treatment +laboratory tests, from 1 to 2 years
Monthly costs of pharmacological treatment of obesity comorbidities (after one year) | 1 year
  Sum of the pharmacological treatment of associated comorbidities (Antidiabetics + Antihypertensives + Statins / lipid-lowering + treatment of hyperuricemia+ Other treatments of obesity comorbidities
Monthly costs of pharmacological treatment of obesity comorbidities (after 2 years) | 2 years
  Sum of the pharmacological treatment of associated comorbidities (Antidiabetics + Antihypertensives + Statins / lipid-lowering + treatment of hyperuricemia+ Other treatments of obesity comorbidities after 2 years
Work absenteeism for 1 year | 1 year
  Number of absences from work (days and hours) due to health problems or medical visits, from baseline from baseline to 1 year
Work absenteeism the second year | 2 years
  Number of absences from work (days and hours) due to health problems or medical visits, from baseline from 1 to 2 years
Body weight loss | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change of body weight from baseline to end of treatment
Waist circumference reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change of Waist circumference from baseline to end of treatment
Blood glucose reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in levels of blood glucose from baseline to the end of treatment
Glycosylated hemoglobin reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in percentage of glycosylated hemoglobin from baseline to the end of treatment
Total cholesterol reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in levels of total cholesterol from baseline to the end of treatment
LDL-cholesterol reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in levels of LDL-cholesterol from baseline to the end of treatment
HDL-cholesterol increase | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in levels of HDL-cholesterol from baseline at the end of treatment
Triglycerides reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in levels of triglycerides from baseline at the end of treatment
Serum uric acid reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in levels of serum uric acid from baseline at the end of treatment
Systolic blood pressure reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in systolic blood pressure from baseline at the end of treatment
Diastolic blood pressure reduction | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in diastolic blood pressure from baseline at the end of treatment
Quality of life (score) | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Change in score in the Short-Form General Health Survey (SF-12) questionnaire from baseline to end of treatment. Raw scores will be calculated as the sum of (re-coded) scale items and transformed to a 0 (negative response) to 100 (positive response) scale. A higher score indicates a better QoL; a positive change (increase in score) in score indicates improvements in QoL while negative change (decrease in score) indicates deterioration.
Number of Participants With Adverse Events | from baseline through treatment completion, an average of 6 months in patients with an initial body mass index of 30 to 35 kg/m2 and an average of 9 months for those patients with initial body mass index higher than 35 kg/m2.
  Number of Participants With Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Rosana Cafardo, Ph, Principal Investigator — Hospital Italiano de Buenos Aires, Argentina; Lucio Criado, Ph, Study Director — Centro Médico Mansilla. Buenos Aires. Argentina
Locations (1):
- Lucio Criado, Buenos Aires, Argentina

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT05833464/Prot_SAP_000.pdf